CLINICAL TRIAL: NCT00784810
Title: A Double-blind, Double-dummy, Parallel Group, Randomised Study to Compare the Efficacy & Tolerability of Oxycodone/Naloxone Prolonged Release (OXN PR) & Codeine/Paracetamol in the Treatment of Moderate to Severe Chronic Low Back Pain or Pain Due to Osteoarthritis
Brief Title: A Study to Compare Oxycodone/Naloxone Prolonged Release Against Codeine/Paracetamol in the Treatment of Moderate to Severe Chronic Low Back Pain or Pain Due to Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Napp Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN4502 (2008-002426-10)
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-09

CONDITIONS: Osteoarthritis; Back Pain
Keywords: Efficacy, tolerability, moderate/severe, oxycodone/naloxone; codeine/paracetamol, chronic low back pain, osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Back Pain; Lymphoma, Follicular | interventions — Oxycodone; Naloxone; acetaminophen, codeine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone/Naloxone Tablets (Experimental): Oxycodone/Naloxone combination
  Interventions: Drug: Oxycodone/Naloxone
- Codeine/Paracetamol Tablets (Active Comparator): Codeine/Paracetamol combination
  Interventions: Drug: Codeine/Paracetamol

INTERVENTIONS:
Drug: Oxycodone/Naloxone — 5/2.5, 10/5 and 20/10 mg oxycodone/naloxone combination, 12 hourly
  Arms: Oxycodone/Naloxone Tablets
Drug: Codeine/Paracetamol — 15/500 and 30/500 mg codeine/paracetamol tablets, 2 tablets 6 hourly
  Arms: Codeine/Paracetamol Tablets

SUMMARY:
The purpose of this study is to compare oxycodone/naloxone combination tablet and codeine/paracetamol tablets in the treatment of moderate to severe chronic low back pain or pain due to osteoarthritis.

DETAILED DESCRIPTION:
This is a randomised, double-blind, double-dummy, parallel group, 12-week study to assess the efficacy and tolerability of oxycodone/naloxone compared to codeine/paracetamol tablets in the treatment of moderate to severe chronic low back pain or moderate to severe pain due to OA of the hip and /or knee.

The screening period will be 3 - 7 days duration. If a subject meets all the screening criteria they may enter the Run-in Period.

During the screening period subjects will continue to take their pre-study pain medication.

The run-in period will be 7 - 14 days duration. During the run-in period subjects will continue to take their pre-study pain medication.

Visit 3 will occur at the end of the Run-in Period (7-14 days after Visit 2). To qualify for entry into the treatment period of the study, subjects must have uncontrolled pain as shown by average daily pain scores of >5 on 4 of the last 7 days of the run in period.

Eligible subjects will be randomised to either oxycodone/naloxone or codeine/paracetamol tablets. Subjects will receive double-blind study medication for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years or older.
2. Female subjects less than one year post-menopausal must have a negative urine pregnancy test recorded prior to the first dose of study medication, be non-lactating, and willing to use adequate and reliable contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectables, combined oral contraceptives, some IUDs, sexual abstinence or vasectomised partner.
3. Subjects with a clinical diagnosis of degenerative or primary OA whose primary pain site is of the hip(s) and/or knee(s) and that require around-the-clock opioid therapy in which the diagnosis may be supported by evidence such as one of the following: MRI, CAT, arthroscopy or x-ray. The clinical imaging of OA may include one or more of the following features: joint space narrowing, degenerative changes, osteophyte formation or subchondral cysts. Subjects will identify the most painful joint (hip or knee) for documentation of OA. Pain measurement will be done at this joint only.
4. Subjects with moderate to severe chronic low back pain e.g osteoarthritis, spinal stenosis, spondylolisthesis, failed back surgery, scoliosis, discogenic disorders such as herniated disc.
5. Subjects who are currently receiving codeine/paracetamol combination tablets up to a maximum dose of 120 mg codeine per day or tramadol up to a maximum dose of 100 mg/day or dihydrocodeine / paracetamol tablets up to a maximum dose of 120 mg dihydrocodeine per day.
6. Subjects willing and able to participate in all aspects of the core study, including use of oral medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, and compliance with protocol requirements as evidenced by providing written, informed consent.
7. Subjects in which the pre-study, non-opioid analgesics, and all other concomitant medications, including those medications for the treatment of depression are anticipated to remain stable throughout the treatment phase of the study.

Exclusion Criteria:

1. Any history of hypersensitivity to oxycodone, naloxone, codeine, ibuprofen, bisacodyl or related products and ingredients.
2. Any contraindication to oxycodone, naloxone, codeine, paracetamol or ibuprofen.
3. Subjects with evidence of significant structural abnormalities of the GI tract (e.g., bowel obstruction, strictures) or any diseases/conditions that affect bowel transit (e.g., ileus, hypothyroidism).
4. Subjects with cancer associated pain.
5. Subjects with secondary osteoarthritis (e.g. fracture, septic, acromegaly etc.).
6. Active alcohol or drug abuse and/or history of opioid abuse.
7. Subjects with Rheumatoid Arthritis.
8. Subjects with non opioid induced constipation.
9. Subjects with evidence of clinically unstable disease, as determined by medical history, clinical laboratory tests, ECG results, and physical examination that, in the investigator's opinion, preclude entry into the study.
10. Subjects with evidence of impaired liver/kidney function upon entry into the study defined as: Aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase levels >3 times the upper limit of normal; Gamma glutamyl transpeptidase ≥5 times the upper limit of normal; Total bilirubin level outside of the reference range unless the value is associated with pre documented Gilbert's Syndrome; Creatinine level outside of the reference range or > 2 mg/dl unless after discussion with the Medical Monitor it is confirmed the subject does not have renal impairment that would preclude the subject's inclusion in the study; In the investigator's opinion the subject has liver and/or kidney impairment to the extent that the subject should not participate in this study.
11. Subjects who have required treatment for the diagnosis of IBS.
12. Subjects receiving hypnotics or other CNS depressants that, in the investigator's opinion, may pose a risk of additional CNS depression with opioid study medication.
13. Subjects with a history of depression or other psychiatric disorder that in the opinion of the investigator is significant enough to exclude the subject from the study.
14. Subjects who are currently involved in legal action regarding their pain condition or subjects in which their pain condition may be of a psychiatric nature.
15. Subjects receiving opioid substitution therapy for opioid addiction (e.g., methadone or buprenorphine).
16. Subjects presently taking, or who have taken naloxone or naltrexone within 30 days of study entry (defined as the start of the Screening Period).
17. Surgery within 2 months prior to the start of the Screening Period, or planned surgery during the12-week treatment period that may affect GI motility or pain levels.
18. Subjects who have received a new chemical entity or an experimental drug within 30 days of study entry (define as the start of the Screening Period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Coventry, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in primary and secondary care in the UK from 6 Feb 2009 to 24 Mar 2010
Pre-assignment Details: 3-7 day screening, following 7-14 day run-in and a 12 week double-blind treatment period.
Groups:
- Oxycodone/Naloxone Tablets (OXN): Oxycodone/Naloxone (OXN) tablets 5,10 and 20 mg
- Codeine/Paracetamol Tablets: Codeine/Paracetamol 15/500 and 30/500 mg
Period: Overall Study
Arm/Group | Oxycodone/Naloxone Tablets (OXN) | Codeine/Paracetamol Tablets
Started | 124 | 123
Completed | 61 | 74
Not Completed | 63 | 49
Not completed — Adverse Event | 32 | 20
Not completed — Lack of Efficacy | 14 | 11
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Administrative | 5 | 8
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone/Naloxone Tablets (OXN) | Codeine/Paracetamol Tablets | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 66 | 70 | 136
  >=65 years | 58 | 53 | 111
Age Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.53) | 63.9 (10.97) | 64.1 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 81 | 158
  Male | 47 | 42 | 89
Region of Enrollment [Number; unit: participants]
  United Kingdom | 124 | 123 | 247

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Pain Score Box Scale-11 (BS-11) Recorded at Week 12 (Average Pain Over Last 24 Hours)
Description: The primary objective was to demonstrate non inferiority of Oxycodone/Naloxone Prolonged Release (OXN PR) compared to codeine/paracetamol in moderate to severe pain as assessed by BS-11 average daily pain scores. The Box Scale-11 is a scale from 0 to 10 (i.e. 0, 1, 2...10), where the subject records their daily pain over the previous 24 hours, by circling the relevant box, where 0 = no pain and 10 = pain as bad as you can imagine. This value is the value recorded at week 12 (average pain over the last 24 hours)
Time Frame: Average daily pain over last 24 hours (at Week 12)
Population: To achieve a study with 80% power at the 1-sided 5% sig level and define non-inferiority to be a relative different less than 1.2. A sample size of 98 subjects per treatment group was required, ie a total of 196 subjects completing the study. The lower number of participants is due to subject withdrawal or lack of data.
Measure: Mean (Standard Deviation); unit: Units on a BS-11 scale at Week 12
Arm/Group | Oxycodone/Naloxone Tablets (OXN) | Codeine/Paracetamol Tablets
Number analyzed (Participants) | 60 | 80
Units on a BS-11 scale at Week 12 | 4.2 (2.139) | 4.64 (2.046)
Statistical Analysis 1: Comparison: Oxycodone/Naloxone Tablets (OXN) vs Codeine/Paracetamol Tablets; To achieve a study with 80% power at the 1-sided 5% significance level, for the purposes of demonstrating non inferiority, a sample size of 98 subjects per treatment group was required, i.e. a total of 196 subjects completing the study; Test type: Non-Inferiority or Equivalence — As above; p = 0.002, Mixed Models Analysis; Mean Difference (Net) = 0.44, 90% CI 1-sided [lower limit -5.65], Standard Error of Mean 1.19

2. Secondary Outcome: Number of Intakes of Rescue Medication (Ibuprofen) Between Visit 8 and Visit 9 for the 2 Groups.
Description: To compare the number of intakes of rescue medication use (ibuprofen) for breakthrough pain between OXN (Oxycodone/Naloxone) and codeine/paracetamol groups. Ibuprofen tablets (400mg up to 3 times per day) were available as rescue medication. This was recorded by the subject in their diary whenever it was taken. The discrepancy in numbers of patients at this stage (between Visit 8 and Visit 9) is due to subject withdrawal during the study. The mean values presented are the "number of intakes of rescue medication" for this period (ie between Visit 8 and Visit 9).
Time Frame: Between visit 8 and 9
Population: The number of participants for analysis is less due to subject withdrawals or lack of data.
Measure: Mean (Standard Deviation); unit: Number of rescue medication intakes
Arm/Group | Oxycodone/Naloxone Tablets (OXN) | Codeine/Paracetamol Tablets
Number analyzed (Participants) | 60 | 80
Number of rescue medication intakes | 13.2 (23.31) | 9.4 (19.94)

ADVERSE EVENTS:
Time Frame: approximately 3 - 4 months, treatment and outcome
Arm/Group | Oxycodone/Naloxone Tablets (OXN) | Codeine/Paracetamol Tablets
Serious Adverse Events (participants affected / at risk) | 3/124 | 4/123
Other Adverse Events (participants affected / at risk) | 27/124 | 32/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone/Naloxone Tablets (OXN) (N=124) | Codeine/Paracetamol Tablets (N=123)
joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
carotid artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
diarrhoea, rectal haemorrhage, abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Head injfury (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Oxycodone/Naloxone Tablets (OXN) (N=124) | Codeine/Paracetamol Tablets (N=123)
Constipation (Gastrointestinal disorders) | 8 | 7
dyspepsia (Gastrointestinal disorders) | 4 | 6
nausea (Gastrointestinal disorders) | 4 | 3
haemorrhoids (Gastrointestinal disorders) | 0 | 4
lower respiratory tract infection (Infections and infestations) | 7 | 4
urinary tract infection (Infections and infestations) | 2 | 5
bronchitis (Infections and infestations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No